CLINICAL TRIAL: NCT06267898
Title: An Observational Audit to Evaluate the Relation Between Transfusions and Iron Toxicity on Major Outcome Parameters in Patients With Adult Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukaemia (CMML) Treated With Myeloablative Conditioning (MAC) and Reduced Intensity Conditioning (RIC) Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT) Without Prior Intensive Antileukemic Therapy by the Chronic Malignancies Working Party by the European Society for Blood and Marrow Transplantation
Brief Title: Non Interventional Study on Iron Toxicity After First Allo-transplant in MDS/CMML
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: EBMT- 842205547
Record Dates: First submitted 2019-08-14; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: MDS; CMML
Keywords: Reduced Intensity conditioning; Myeloablative conditioning; Allogeneic stem cell transplantation; iron toxicity; Non-interventional; Observational study; MDS; CMML

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Stem cell transplantation and blood product transfusions are standard of care for Myelodysplastic Syndromes (MDS). Several studies have shown changes in serum ferritin and non-transferrin-bound iron (NTBI) in patients undergoing stem cell transplantation. A large proportion of MDS patients are at risk for organ damage from tissue siderosis, due to the development of iron overload.

Toxic effects of iron may play an important role in the complications associated with HSCT. Iron chelation therapy may reduce the acute and chronic treatment-related toxicity by removing excess of iron, iron radicals and reactive oxygen species (ROS).

There is little information about the efficacy and safety of iron chelation in MDS patients. This audit wants to evaluate the effect of iron toxicity on treatment-related mortality in untreated, adult MDS or CMML patients during and after treatment with myeloablative conditioning (MAC) and reduced intensity conditioning (RIC) allo-HSCT, by prospectively collecting data from 200 MDS or CMML patients from 2009 onwards.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To evaluate in adult MDS or CMML patients the correlation between iron toxicity and treatment-related mortality in the context of the treatment of such toxicity with iron chelation during and after treatment with allo-HSCT

DETAILED DESCRIPTION:

Myelodysplastic syndromes (MDS) form a complex and heterogeneous group of bone marrow failure disorders. These are characterized by ineffective hematopoiesis leading to peripheral cytopenias and morphologic dysplasia. The incidence of MDS is about 5 per 100,000 persons a year in the general population. After 60 years of age the incidence increases tot 20-50 per 100,000 persons a year.

Care for MDS includes amelioration of hematological deficits with blood product transfusions, and stem cell transplantation after a standard myeloablative regimen. At the moment stem cell transplantation is the only known curative treatment for MDS patients . Allogeneic Stem cell transplantation can lead to considerable treatment-related morbidity and mortality among patients. Insight in factors contributing to treatment related mortality, could lead to a better treatment regimen in patients who are treated with allo-HSCT and subsequently lead to overall lower treatment related mortality.

Red blood cell transfusion therapy is used to prevent anemia-related morbidity, and to improve quality of life. However, non-transfusion dependent patients have a significantly better prognosis than transfusion dependent patients.

The increased mortality of transfused patients can partly be attributed to iron overload. Iron overload is a common acute and long-term event associated with autologous and allogeneic hematopoietic stem cell transplantation (HSCT). The main cause of iron overload is chronic transfusion therapy. Frequent blood transfusions lead to an increase in ferritin levels, transferrin saturation and in the appearance of non-transferrin-bound iron (NTBI). Iron overload is also observed in non-transfused patients with MDS. This may be due to the release of toxic iron radicals by the intensive treatment itself and its associated ineffective hematopoiesis, and some other less well defined processes. Ineffective hematopoiesis for example, either a feature of the underlying disease or a consequence of the intensive treatment, leads to growth and differentiation factor (GDF-15) over-expression which inhibits the production of hepcidin in the liver. This leads to increased iron absorption and increased iron toxicity.

When the acute storage capacity for body iron is exceeded, organs, such as liver, heart and endocrine glands, are loaded with free iron. This leads to free radical generation, tissue damage, and subsequently organ dysfunction.

Individuals with IPSS lower-risk disease or high-risk patients who respond favorably to intensive antileukemic therapy, may survive long enough to develop clinical consequences of iron overload. An increased iron load leads to toxic and infectious events even during the first 3 months after transplantation.

Several different investigations are useful to determine iron overload. These include imaging of liver and heart, tissue histology, and serum ferritin, transferrin saturation and non-transferrin-bound iron (NTBI). Accuracy of imaging studies and feasibility of standard tissue histology has been questioned. Serum ferritin and NTBI levels are widely used to quantify iron overload, but are also limited in their use. Ferritin is elevated in various inflammatory situations, as well as in hepatic damage. Therefore one should always be careful in interpreting serum ferritin variations. When combined with liver enzymes and inflammation markers, such as fibrinogen and C-reactive protein (CRP), ferritin, transferrin saturation and NTBI levels can be used as a simple (and non-invasive) diagnostic step to determine iron overload.

Although chronic red blood cell transfusions leading to iron overload are common among patients with MDS, the clinical implications and the value of iron chelation therapy in MDS remain unclear. Iron chelation therapy could improve the survival in transfusion-dependent MDS patients, by removing excess iron, iron radicals and reactive oxygen species (ROS). This may lead to a reduction in acute and chronic treatment-related toxicity and a reduction in treatment-related mortality.

Results with iron chelation are mostly gained in studies which have been performed in other transfusion dependent diseases, like thalassemia. It is often stated that the survival rate in MDS is too low, due to coexisting morbidity and that the MDS patients are too old to benefit from chelation therapy. However, patients with MDS could be more vulnerable to the toxic effects of iron overload and therefore benefit more from iron chelation therapy in a shorter period.

The recent development of oral iron chelators, like deferasirox and deferiprone, might lead to a breakthrough in chelation therapy for MDS patients. Although most information stems from trials performed on non-MDS patients, oral chelators promise to be effective and convenient alternatives for subcutaneously administered iron chelators, like desferoxamine. The biggest benefit of these drugs is their oral use. Continuous subcutaneous infusions are inconvenient and may be associated with local side effects. On the other hand, both deferiprone and deferasirox can also produce relevant side effects.

There is very little literature available to guide recommendations for management and treatment of iron overload in patients with low-risk MDS. Most information about iron overload and chelation stems from non-MDS patients. More studies are needed to quantify effects of iron overload in MDS patients and to determine efficacy and safety of oral chelators over other therapies. This international observational audit will provide insight in correlation between iron overload and outcome of disease in MDS or CMML patients.

An ongoing retrospective analysis by the MDS subcommittee of the EBMT-CLWP showed that the number of transfusions administered prior to the allogeneic SCT had a significant impact on survival by a reduced non relapse mortality in patients who received less than 20 units prior to the transplantation. Pre-transplantation ferritin levels were only reported in a minority of the patients, but also ferritin levels appear to influence the non relapse mortality in this group of patients (personal communication). Therefore, the proposed international observational audit will provide insight in correlation between iron overload and outcome of disease in MDS or CMML patients.

RESEARCH DESIGN:

Centers will be asked to register prospectively patients in this observational, non-interventional audit. Patients will be treated according to local protocols. Both Myelo-ablative conditioning (MAC) and Reduced Intensity Conditioning (RIC) are allowed.

It is advised to treat iron overload from 2 months after allogeneic HSCT onwards if serum ferritin levels are over 1,000 g/l. Both phlebotomies and iron chelation therapy are assumed to be a policy of the center applicable to all patients treated by that center; each center is required to accurately state its "intention-to-treat" policy, i.e. under what conditions a decision for phlebotomy and/or iron chelation therapy is normally reached (although centers are allowed to deviate from this general policy if deemed necessary),based on individual patient or physician preference. This "Intention-to-treat-policy" should be given before inclusion of the first patient in this observational audit. Details of the chelation and the phlebotomy therapy can be found on the Website of the EBMT (details: http://www.ebmt.org/ClinicalTrials/observational audits/ not available yet).

Data will be collected by forms or files based on existing MED-B forms and an additional questionnaire.

Follow-up data will be collected at 3 months, 6 months and every 6 months thereafter

STUDY POPULATION:

200 adult patients with cytologically proven untreated MDS or CMML, according to the FAB or the WHO classification, transplanted with myeloablative or reduced intensity conditioning allo-HSCT from May 2009 onwards.

RESEARCH VARIABLES

* Patients' features
* Centres' features
* Initial diagnosis
* Interval between diagnosis and HSCT
* Subclassification and status of disease at HSCT
* Complications: liver (transaminases, bilirubin, incidence VOD), kidney impairment, infections
* Additional therapies
* Relapse or progression
* Last disease and patient status
* Donor
* Transplantation
* Graft manipulation
* Engraftment
* Comorbid conditions
* Preparative treatment
* Graft versus Host disease
* RBC transfusions before and after transplantation
* Ferritin levels, CRP, transferrin saturation, NTBI
* Chelation therapy: start therapy and average daily dosage per month
* Phlebotomy therapy: start therapy and average number of phlebotomies per month
* Follow up

ANALYSIS The primary outcome of this audit is non-relapse mortality (treatment related mortality).

Secondary outcomes are treatment-related toxic effects, relapse rate, event-free survival and overall survival.

Variables to be analyzed for their predictive ability on the above mentioned outcome variables, are:

* Transfusion dependency, number of transfusions, hemoglobin levels
* ferritin levels, transferrin saturation, C-reactive protein (CRP)
* iron chelation therapy (prior and postSCT)
* phlebotomy therapy
* disease classification at SCT
* age patient,
* donor type
* female-donor/male recipient vs other combinations
* SCT conditioning type
* interval diagnosis and SCT, cytogenetics
* T-cell depletion
* acute and chronic GVHD
* length of survival
* primary causes of death
* relapse and complications

METHOD OF ANALYSIS:

For the primary objective(s), non-relapse mortality and relapse incidence will be analyzed together in a competing risk framework, based on cause-specific hazard estimates stemming from the appropriate Cox models.

The center will be introduced as a random effect. Since this is an observational and not a randomized study, comparison of treatment policies with respect to outcome is difficult due to the interplay of treatment policy and the actual occurrence of toxicity and a possible center effect. Hence the prudent way to proceed is a thorough analysis within the subgroups based on the center policy (the actual application of a specific treatment is depending on center policy rather than the individual characteristics of the patient, so the covariate "iron toxicity therapy" will be used as a intention-to-treat stratification factor rather than a covariate).

The influence of iron toxicity in its broadest sense on the primary outcome variables is studied by taking iron toxicity parameters as an additional covariate in a full Cox model for non-relapse mortality as well as relapse incidence using known predictors for these outcomes among MDS or CMML patients.

The entire analysis will be a careful evaluation of the above mentioned parameters in an observational context and therefore a detailed statistical plan listing all possible hypotheses to be tested, is not provided a priori since the observational nature of this audit will most likely induce hypothesis generating statements rather than hypothesis testing ones.

The methodology applied can however be stated in advance. Apart from Cox regression models and a competing risk framework, the data will be analyzed according to the repeated measurements structure induced by the repeated observations. In particular the predictive ability of toxicity measures on any variables occurring later in time (whether events or other continuous measures) will be studied in the context of mixed models, accounting for center effects. These analyses focus on prediction of parameters at 3 months after SCT, 1 year after SCT, and 2 years after SCT. An interim analysis will be performed at the time point when the first 100 patients have a follow-up of one year after SCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MDS or CMML, according to FAB-criteria (RA, RARS, RAEB, RAEBt, CMML) or according to WHO-criteria (RA, RARS, RAEB-1, RAEB-2, RCMD, RCMD-RS, with isolated del(5q), MDS OR CMML-U)
* Patients with transformed MDS or CMML to AML at time of transplant
* Patients received myeloablative or RIC allo-HSCT as primary treatment
* Diagnosis at time of transplant
* Informed Consent and of legal age at the time of obtaining informed consent (18+)
* ECOG performance status 0-2

Exclusion Criteria:

* Patients with previous intensive antileukemic therapy (intensive chemotherapy and/or HSCT); previous treatment with immunomodulatory drugs (thalidomide, or lenalidomide) or hypomethylating agents (Vidaza, decitabine) is allowed
* Patients with juvenile chronic myelomonocytic leukemia (jMML)
* Patients with secondary or therapy-related AML and MDS or CMML after treatment with immunosuppressive or cytotoxic treatment for a nonmyeloid malignancy
* Patients who received auto-HSCT
* Candidates for cord blood HSCT or syngeneic HSCT
* Inadequate renal function (ECC <60 ml/min and/or creatinine >2.5 times upper limit of normal value)
* Inadequate hepatic function (transaminases >2.5 times upper limit of normal value)
* History of seizures
* Pregnancy and women of child-bearing potential and not using adequate contraceptives
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: eligible patient from EBMT centres
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2015-05-21 (Actual)

PRIMARY OUTCOMES:
non-relapse mortality (treatment related mortality). | 2 years after HSCT

SECONDARY OUTCOMES:
treatment-related toxic effects | 2 years after HSCT
relapse rate | 2 years after HSCT
event-free survival | 2 years after HSCT
overall survival | 2 years after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: T. de Witte, MD, Principal Investigator — Radboud University Medical Center; E. Cremers, Principal Investigator — VUMC - VU University Medical Centre Amsterdam; N. Kröger, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (6):
- Belgium (3):
  - Antwerp University Hospital (UZA), Antwerp
  - University Hospital Gasthuisberg, Leuven
  - University of Liege, Liège
- Charles University Hospital, Pilsen, Czechia
- Germany (2):
  - University Hospital, Essen
  - University Hospital Leipzig, Leipzig